CLINICAL TRIAL: NCT01881880
Title: Value of Tomosynthesis in Breast Lesion Characterization and Breast Cancer Staging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8904
Record Dates: First submitted 2013-03-22; First posted 2013-06-20 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: Tomosynthesis; Mammography; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tomosynthesis (Other): Bilateral mammography with 4 views Tomosynthesis
  Interventions: Device: Bilateral mammography with Tomosynthesis

INTERVENTIONS:
Device: Bilateral mammography with Tomosynthesis — no intervention pre specified to be administered to participants

SUMMARY:
Study Rationale: an accurate breast cancer staging has a great impact in the management of a breast cancer. MRI is considered as the most sensible exam for this staging. However it has a low specificity and it may result in extra testing and stress for the patient, add to costs, and delay treatment. By contrast, Tomosynthesis is performed during the same time than mammography and has a good specificity. Although this modality is very promising, it has not been assessed in a population of consecutive patients.

Study objectives: To compare the diagnostic performance of preoperative bilateral Combo mode (MG+Tomosynthesis) versus mammography among women with breast cancer for the detection of additional multifocal, multicentric, and contralateral cancers.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 40 years old
* Subject with a new lesion recommended for biopsy, whatever the modality which detected the lesion (clinical examination, mammography, tomosynthesis, US, or MRI)

Exclusion Criteria:

* Subjects with BRCA mutation or at high genetic risk
* Subjects who have breast implants
* Personal history of breast cancer
* Subjects who are pregnant or who think they may be pregnant
* Subjects who are breast-feeding
* Subjects who are unable or unwilling to tolerate study constraints
* Subjects unable or unwilling to undergo informed consent
* Subject with no rights from the national health insurance programme

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
diagnostic performance of preoperative bilateral Combo mode (MG+Tomosynthesis) versus mammography among women with breast cancer for the detection of additional multifocal, multicentric, and contralateral cancers. | 1 year
  In all sites, Mammography and Tomosynthesis will be standardised and performed according to the Combo mode with 2 views for each breast.
  Any additional breast lesion assigned a BI-RAD 4 or 5 score after the full staging work-up will be biopsied under the best imaging method.
  (BIRADS scale : BIRADS 4a or higher is considered to be positive for cancer )
  The Gold Standard diagnosis is defined as the final diagnosis at 1 year on the basis of the most severe histopathologic result (surgery, biopsy) for that lesion.
  A retrospective imaging evaluation of mammography versus Combo mode will be performed for the patients diagnosed with a breast cancer lesion. This retrospective imaging evaluation will be conducted centrally within the assessment committee at the lesion, breast and patient level.

SECONDARY OUTCOMES:
performance of MG vs Combo (MG+Tomosynthesis) for the diagnosis of multicentricity | 1 year
  Concerning breasts lesions : assessing multicentricity by MG and Combo for the presence of one BI-RADS 4-5 lesions, presence of multifocal BI-RADS 4-5 lesions presence of multicentric BI-RADS 4-5 lesions
  A retrospective imaging evaluation of mammography versus Combo mode will be performed for the patients diagnosed with a breast cancer lesion. This retrospective imaging evaluation will be conducted centrally within the assessment committee at the lesion.
performance of MG vs Combo (MG+Tomosynthesis) for the diagnosis of multifocality | 1 year
  concerning Breasts lesions : assessing multifocality by MG and Combo for the presence of one BI-RADS 4-5 lesions, presence of multifocal BI-RADS 4-5 lesions presence of multicentric BI-RADS 4-5 lesions
  A retrospective imaging evaluation of mammography versus Combo mode will be performed for the patients diagnosed with a breast cancer lesion. This retrospective imaging evaluation will be conducted centrally within the assessment committee at the lesion, breast and patient level.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Taourel, Principal Investigator — UH Montpellier
Locations (6):
- France (6):
  - Private Hospital oh Antony, Antony
  - UH Grenoble, Grenoble
  - Oscar Lambret Center, Lille
  - Jean Mermoz Hospital, Lyon
  - UH Montpellier, Montpellier
  - Hospital Valenciennes, Valenciennes

REFERENCES:
- [Derived] Fontaine M, Tourasse C, Pages E, Laurent N, Laffargue G, Millet I, Molinari N, Taourel P. Local Tumor Staging of Breast Cancer: Digital Mammography versus Digital Mammography Plus Tomosynthesis. Radiology. 2019 Jun;291(3):594-603. doi: 10.1148/radiol.2019182457. Epub 2019 Apr 9. PMID 30964425